CLINICAL TRIAL: NCT01541683
Title: The Effect of Mentholyptus Drops (Halls®) on the Palatability of PEG-Electrolyte Solution (FORTRANS®) in Colonoscopy Preparation: A Randomized Controlled Trial
Brief Title: The Effect of Mentholyptus Drops on the Palatability of PEG-Electrolyte Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ala'a Sharara, Head and Professor, Division of Gastroenterology and Hepatology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IM.AS1.28
Record Dates: First submitted 2012-02-21; First posted 2012-03-01 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Colon Cancer
Keywords: PEG-electrolyte solution; bowel cleansing; Mentholyptus drops; Palatability
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Halls (Experimental): every patient will drink 4 Liters of PEG solution (FORTRANS®) split into 2 days with sugar-free mentholyptus drops (2 L at 7-9 pm on the day prior to the colonoscopy with Halls®, and 2 L on the day of the colonoscopy to be completed a minimum of 1.5 hours before the procedure with Halls®).
  Interventions: Other: PEG solution (Fortrans®) and Mentholyptus Drops (Halls®)
- no Halls (Other): Every patient will drink 4 liters of PEG solution (FORTRANS®) split into 2 days (2 L at 7-9 pm on the day prior to the colonoscopy, and 2 L on the day of the colonoscopy to be completed a minimum of 1.5 hours before the procedure)
  Interventions: Other: PEG solution (Fortrans®)

INTERVENTIONS:
Other: PEG solution (Fortrans®) and Mentholyptus Drops (Halls®) — Patients will be instructed to drink 4 Liters of PEG solution (FORTRANS®) split into 2 days while sucking on sugar-free mentholyptus drops (2 L at 7-9 pm on the day prior to the colonoscopy while continuously sucking on Halls®, and 2 L on the day of the colonoscopy to be completed a minimum of 1.5 hours before the procedure while continuously sucking on Halls®)
  Arms: Halls
Other: PEG solution (Fortrans®) — 4 liters of PEG solution (FORTRANS®) split into 2 days (2 L at 7-9 pm on the day prior to the colonoscopy, and 2 L on the day of the colonoscopy to be completed a minimum of 1.5 hours before the procedure)
  Arms: no Halls

SUMMARY:
The investigators aim is to study the efficacy of mentholyptus drops in improving the palatability of PEG-electrolyte solution used in bowel cleansing for colonoscopy. The study is a randomized controlled trial which will include patients undergoing elective colonoscopy at the American University of Beirut Medical Center. Patients will be randomized into one of two study arms using a computer generated randomization list. Patients assigned to the intervention arm will be asked to have candy (Halls®) during the whole 2 hours period while drinking the PEG solution unlike the control arm patients who will only receive the PEG solution. All patients will then be evaluated for the tolerability of the preparation while taking into account the palatability of the solution as main outcome and the remaining volume of the PEG solution and side effects as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* elective colonoscopy
* consent to the study

Exclusion Criteria:

* pregnant or lactating women
* age less than 18 years
* significant gastroparesis
* gastric outlet obstruction
* ileus
* known or suspected bowel obstruction or perforation
* phenylketonuria
* glucose-6-phosphate dehydrogenase deficiency
* severe chronic renal failure (creatinine clearance <30 mL/minute)
* severe congestive heart failure (NYHA class III or IV)
* dehydration
* severe acute inflammatory disease
* compromised swallowing reflex or mental status
* uncontrolled hypertension (systolic blood pressure ≥170 mm Hg, diastolic blood pressure ≥100 mm Hg)
* toxic colitis or megacolon
* previous colonoscopy within the last 5 years
* active Inflammatory bowel disease
* previous colectomy or partial colectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
measurement of Palatability of the PEG-electrolyte solution | 1.5 hours after drinking the solution
  patients will be asked to assess the palatability of the colon preparation solution (Fortrans®) by giving it a score on a scale from 1 to 5 with 1 being disgusting and 5 being tasty after drinking the whole solution and immediately prior to the colonoscopy

SECONDARY OUTCOMES:
volume remaining of the colon preparation solution | 1.5 hours after drinking the solution
  Patients will be asked to bring with them to the endoscopy suit the volume remaining, if any, of the colon preparation solution that they were not able to drink. The volume remaining will be measured by the research fellow using a graduated cylinder.
Side effects | 1.5 hours after drinking the solution
  number of patients who experienced nausea, vomiting, bloating, abdominal cramps or headaches while drinking the solution.

CONTACTS AND LOCATIONS:
Overall Officials: Ala I Sharara, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Beyrouth, Lebanon

REFERENCES:
- [Derived] Sharara AI, El-Halabi MM, Abou Fadel CG, Sarkis FS. Sugar-free menthol candy drops improve the palatability and bowel cleansing effect of polyethylene glycol electrolyte solution. Gastrointest Endosc. 2013 Dec;78(6):886-891. doi: 10.1016/j.gie.2013.05.015. Epub 2013 Jun 13. PMID 23769143